CLINICAL TRIAL: NCT05990114
Title: Evaluation of the Effect of Structured Caregiver Support Program on the Levels of Care Burden, Psychological Well-Being and Psychological Resilience of Informal Caregivers of Alzheimer's Patients
Brief Title: Evaluation of the Structured Caregiver Support Program (SCSP) in Terms of Various Parameters
Acronym: SCSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Hande Kirisik, Lecturer, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: KAEK-28
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease
Keywords: psychosocial intervention; Alzheimer's disease; caregivers; care burden; psychological well-being; psychological resilience
MeSH Terms: conditions — Alzheimer Disease; Caregiver Burden; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The structured caregiver support program is a psychosocial training program developed to improve caregivers' burden of care, psychological well-being and resilience.This training program will be applied to the intervention group.
  Interventions: Other: The structured caregiver support program
- control group (No Intervention): No intervention will be applied to the control group.

INTERVENTIONS:
Other: The structured caregiver support program — It consists of 8 sessions in total. It is planned as once a week and 45 minutes.
  Arms: intervention group

SUMMARY:
The aim of this clinical study is to examine the effect of an intervention program developed for informal caregivers of Alzheimer's patients on caregivers' burden of care, psychological well-being and psychological resilience.The main questions it aims to answer are:

1. What is the effect of the Structured Caregiver Support Program (SCSP) on caregivers burden?
2. What is the effect of the SCSP on psychological well-being?
3. What is the effect of the SCSP on psychological resilience?

Participants (intervention group) will attend at least 6 sessions of an 8-session SCSP.

Researchers will compare with the control group to see if the training provided is effective.

DETAILED DESCRIPTION:
People around the world are now living longer. The number of elderly people in need of care is increasing, especially among the population aged 80 and over, which is defined as advanced old age. Elderly care in Turkey is largely informal by family members. A significant proportion of caregivers suffer from the burden of care. Alzheimer's disease (AD) is a neurodegenerative and progressive disease that causes need for care in advanced age. Caregivers of people with AD report more stress, burden and depression than caregivers of other patients, especially in cases where neuropsychiatric symptoms are evident. Psychological well-being and psychological resilience of caregivers are also negatively affected by the care process. Therefore, caregivers need psychological and social support. The aim of this study is to evaluate the effect of the Structured Caregiver Support Program, which will be created to support caregivers psychologically and socially, on the caregiving burden, psychological well-being and psychological resilience levels of informal caregivers caring for Alzheimer's patients.

Mixed design consisting of quantitative and qualitative research methods will be used in the research.The quantitative dimension of the research will be carried out as a randomized controlled experimental study and a pre-test and post-test order will be used.In this context, an intervention program was created to examine the effect of the Structured Caregiver Support Program on caregivers' burden of caregiving, psychological well-being and psychological resilience.There will be two different groups in the study, namely the intervention group and the control group. The trial is designed as a group intervention. Therefore, all 25 caregivers in the intervention group will attend the sessions at the same time. Participants who volunteer to participate in the study will be randomly assigned to the intervention and control groups.SCSP intervention will be applied to the intervention group and no intervention will be applied to the control group.Pre-test and post-test will be applied to both the intervention and control groups before and after the intervention program.

The universe of the research consists of caregivers of patients with Alzheimer's diagnosis followed up in the Alzheimer's Social Life Center of a municipality in Ankara between September and November 2023.The sample of the study consists of caregivers who meet the criteria for inclusion in the sample of patients with Alzheimer's diagnosis followed in the Alzheimer's Social Life Center of a municipality in Ankara between September and November 2023.

ELIGIBILITY:
Inclusion Criteria:

* Providing informal care to an individual with mild or moderate Alzheimer's disease
* Being a primary caregiver
* Having been caring for the patient for at least 6 months
* Providing care to the patient for at least 6 hours a day
* The caregiver is 18 years or older
* Residency of the caregiver in the province of Ankara
* Willingness and volunteering to participate in the research

Exclusion Criteria:

* Hearing and understanding difficulties
* Having a psychiatric disorder
* Receiving any therapy services
* Caregivers who did not attend two or more of the eight interviews were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Zarit Burden Interview | change from baseline to the end of the 8th week
  This scale, which was developed by Zarit, Reever and Bach-Peterson in 1980, is used to measure the stress of caregivers.A minimum of 0 and a maximum of 88 points can be obtained from the scale. A high score on the scale indicates a high level of distress.

SECONDARY OUTCOMES:
Psychological Well-Being Scale | change from baseline to the end of the 8th week
  The 8-item Psychological Well-Being Scale, developed by Diener et al. in 2009, includes important elements of human functioning such as positive relationships, feelings of efficacy, and having a meaningful and purposeful life, and evaluates the individual's psychological well-being.A minimum of 8 and a maximum of 56 points can be obtained from the scale. A high score indicates that the person has many psychological resources and strengths.
Brief Resilience Scale | change from baseline to the end of the 8th week
  It is a 6-item self-report scale developed by Smith et al. in 2008. After the reverse coded items in the scale were translated, high scores indicate high psychological resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Hande Kirisik, Lecturer, Principal Investigator — Ankara University
Locations (1):
- Akdeniz University, Antalya, Konyaaltı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No